CLINICAL TRIAL: NCT07124260
Title: Dysbiosis of Gut-Tongue Coating Microbiota Crosstalk and Its Clinical Association With Diminished Ovarian Reserve: A Microbiome-Based Case-Control Study
Brief Title: Characterization of Gut and Tongue Coating Microbiota in Patients With Diminished Ovarian Reserve
Acronym: CGTCMPDOR
Status: Recruiting | Type: Observational
Sponsor: Hangzhou TCM Hospital Affiliated to Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Wenjun Xiao, gynecologist, Hangzhou TCM Hospital Affiliated to Zhejiang Chinese Medical University
Other Study IDs: DOR CDJQ STJQ case control
Record Dates: First submitted 2025-08-01; First posted 2025-08-15 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Diminished Ovarian Reserve
MeSH Terms: interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The preserved biological samples comprised fresh human fecal specimens and human tongue coating samples.
  Microbial DNA will be extracted from fecal and tongue coating samples using the QIAamp DNA Microbiome Kit (Qiagen, Hilden, Germany). Whole-genome DNA was isolated via the centrifugal adsorption column method, and DNA quality was evaluated by agarose gel electrophoresis (1.0% agarose concentration, 150V voltage, 20-minute electrophoresis time). Samples meeting the following criteria-distinct genomic bands, total DNA quantity >200 ng, DNA concentration >10 ng/μL, OD260/280 >1, and OD260/230 >2-were selected for sequencing library construction and subsequent sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diminished Ovarian Reserve Group
  Interventions: Diagnostic Test: gut microbiota; Diagnostic Test: tongue coating microbiota; Diagnostic Test: tongue picture
- Healthy Control Group
  Interventions: Diagnostic Test: gut microbiota; Diagnostic Test: tongue coating microbiota; Diagnostic Test: tongue picture

INTERVENTIONS:
Diagnostic Test: gut microbiota — Fresh fecal samples were collected from patients during the non-menstrual period and subjected to 16S rDNA sequencing.
Diagnostic Test: tongue coating microbiota — Tongue coating samples were collected under fasting conditions between 6:00-9:00 AM on the same day as fecal specimen collection and subjected to 16S rDNA sequencing.
Diagnostic Test: tongue picture — Tongue images were captured under fasting conditions between 6:00-9:00 AM on the same morning as fecal specimen collection.

SUMMARY:
The goal of this observational study is to investigate the distinct tongue manifestation characteristics in patients with diminished ovarian reserve (DOR) compared to healthy individuals, and to clarify the features of tongue coating microbiota, gut microbiota, and their interrelationships in DOR patients. The main question it aims to answer is:

Whether there are significant differences in tongue manifestations, tongue coating microbiota, and gut microbiota characteristics between DOR patients and healthy populations; Whether associations exist between tongue coating microbiota and gut microbiota in DOR patients; Whether the pathogenesis of DOR may influence estrogen metabolism through alterations in oral and gut microbiota.

DETAILED DESCRIPTION:
This study enrolled DOR patients and healthy women as controls to systematically analyze compositional differences in intestinal and tongue coating microbiota between the two groups. Using 16S rDNA sequencing technology combined with bioinformatics methods, we screened characteristic microbiota associated with DOR and identified microbial markers significantly correlated with serum estrogen levels (AMH, FSH) through Spearman correlation analysis. We further compared abundance differences of homologous bacteria between tongue coating and gut microbiota to determine whether DOR alters the abundance or prevalence of specific bacterial species by affecting tongue-gut axis microbial interactions. The potential of tongue-gut differential microbiota combinations as non-invasive diagnostic biomarkers for DOR was explored.

ELIGIBILITY:
Inclusion Criteria Developed in accordance with:

The 13th Five-Year Plan textbook Obstetrics and Gynecology (9th Edition) by China National Health Commission The 14th Five-Year Plan National Key Publication Reproductive Endocrinology (2nd Edition) Expert Consensus on Clinical Diagnosis and Treatment of Diminished Ovarian Reserve (2022)

Inclusion Criteria:

* Female patients aged >20 years.
* Diagnosis required meeting the essential criterion of AMH <1.1 ng/mL plus at least one supportive criterion: FSH >10 IU/L, FSH/LH ratio >3.0, or AFC <5-7 follicles (measured on menstrual days 2-3).
* Conscious with intact cognitive/linguistic functions to comply with study protocols.
* Approved by Ethics Committee of Hangzhou TCM Hospital Affiliated to Zhejiang Chinese Medical University, with written informed consent obtained.

Exclusion Criteria:

* Female participants aged <20 years.
* Women in menopause, pregnancy, or lactation period.
* Participants with comorbidities that may interfere with drug efficacy (e.g., severe chronic diseases).
* Severe primary disorders involving cardiovascular, hepatic, renal, hematopoietic systems, or psychiatric illnesses.
* Non-compliance with medication protocols during the study, or cases with undeterminable efficacy outcomes/incomplete data.
* Use of sex hormone therapy within the past 3 months.
* Diagnosis of reproductive system malignancies.
* Gastrointestinal disorders or abnormal liver function.
* Poor adherence to study protocols or lost to follow-up.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender woman
Study Population: Women with diminished ovarian reserve
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Follicle stimulating hormone | On day 2 or 3 of the menstrual phase during the first menstrual cycle following participant enrollment.
  Follicle stimulating hormone in IU/L

SECONDARY OUTCOMES:
anti-mullerian hormone | On the first day following participant enrollment.
  Anti-mullerian hormone in ng/mL
Antral Follicle Counting | On day 2 or 3 of the menstrual phase during the first menstrual cycle following participant enrollment.
  The antral follicle counting will be performed via transvaginal ultrasound with the patient in the lithotomy position after bladder voiding. The total number of antral follicles measuring 2-6 mm in diameter within both ovaries will be recorded and reported as individual counts.
gut microbiota | Fresh fecal samples were collected in the morning under fasting conditions within one week after menstruation completion during the first menstrual cycle following enrollment.
  Fecal midstream samples (≤10g) were collected using sterile sampling kits, immediately flash-frozen in liquid nitrogen, and stored at -80℃. Gut microbiota profiling was performed via 16S rRNA gene sequencing for both the Healthy Control Group and Diminished Ovarian Reserve Group. Differential gut microbiota at genus-level and higher taxonomic ranks between groups will be reported.
tongue coating microbiota | Tongue coating samples were collected in the morning under fasting conditions within one week after menstruation completion during the first menstrual cycle following enrollment, with priority given to coordinating collection on the same day as fecal spe
  Researchers collected tongue coating samples using sterile tongue swabs with 10 rotational scrapes at the mid-tongue region. Specimens were immediately flash-frozen in liquid nitrogen and stored at -80℃. Tongue microbiota profiling was performed via 16S rRNA gene sequencing for both the Healthy Control Group and Diminished Ovarian Reserve Group. Differential microbial communities at genus-level and higher taxonomic ranks between groups will be reported.
pregnancy outcome | 1-year follow-up period post-detection
  In this context, pregnancy outcome specifically refers to term delivery status. All participants underwent systematic follow-up through telephone interviews or medical record retrieval to document the number of subjects achieving term delivery in both study cohorts.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou TCM Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data may be available upon reasonable request to the Ethics Committee, subject to a data transfer agreement.